CLINICAL TRIAL: NCT05485350
Title: A Single-arm Clinical Study of Anlotinib Combined With Penpulimab Plus SBRT in Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Anlotinib , Penpulimab Combined With SBRT for Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L056
Record Dates: First submitted 2022-07-09; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib combined with SBRT and penpulimab (Experimental)
  Interventions: Drug: Anlotinib Hydrochloride; Drug: penpulimab; Radiation: SBRT

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — 12 mg/d, d1-14, q3w
  Other Names: AL3818; Anlotinib Hydrochloride Capsules; FuKeWei
Drug: penpulimab — 200mg, ivgtt, d1, q3w
  Other Names: AK105
Radiation: SBRT — 55-180Gy

SUMMARY:
This study will explore the effectiveness and safety of the combination therapy of anlotinib , penpulimab and SBRT in patients with metastatic non-small Cell Lung Cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, no gender limit；
* Histological or cytological diagnosis of stage IV non-small cell lung cancer（NSCLC）
* The patients joined the study voluntarily and signed an informed consent form (ICF). They had good compliance and cooperated with follow-up.
* Patients with advanced NSCLC who have received one or two systemic treatments, and those who are unwilling to accept or cannot tolerate systemic chemotherapy can also be enrolled. If it is a driver gene mutation-positive (EGFR, ALK) patient, it must be accepted after receiving the corresponding targeted therapy resistance or intolerable toxicity, No secondary susceptible mutations were eligible for enrollment.
* Has at least five disseminated lesions for SBRT , and measurable lesion that meets the RECISTv1.1 standard。
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
* The expected survival time ≥ 3 months;
* The functions of important organs meet the following requirements (no blood components and cell growth factors are allowed to be used 2 weeks before the start of the research treatment): Absolute Neutrophil Count (ANC) ≥1.5×10 E+9/L, Hemoglobin (HB) ≥9g/dL, Platelets (PLT)≥90×10 E+9/L, Serum Albumin (ALB)≥2.8g/dL, Total Bilirubin (TBIL) ≤1.5 ULN, ALT、AST≤2.5 UILN(If abnormal liver function is caused by liver metastasis, ≤5 ULN), Serum creatinine sCr≤1.5 ULN, endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula) , Normal thyroid function;
* For female subjects of childbearing potential, a serum pregnancy test should be performed within 7 days prior to the administration of the first study intervention (study drug, radiation therapy) and have a negative result. Subjects are required to agree to use highly effective contraception and continue until at least 120 days after discontinuation of trial treatment

Exclusion Criteria:

* The lesion has received prior radiotherapy and is not suitable for SBRT;
* Currently participating in interventional clinical research and treatment, or receiving other research drugs or treatment with research equipment within 4 weeks before the first administration;
* Imaging (CT or MRI) shows evidence of tumour invasion of large blood vessels or poorly demarcated blood vessels or the presence of cavities and necrotic lesions in the lungs；
* With active bleeding or perforation or a hereditary or acquired bleeding tendency present, with a daily haemoptysis of ≥2.5mL in the 3 months prior to screening.
* Suffer from active autoimmune diseases that require hormone or immunomodulatory treatment;
* Have received anti-tumor monoclonal antibodies (mAb) within 4 weeks before using the study drug for the first time, or the adverse events caused by the previously received drug have not recovered (ie ≤ grade 1 or reached the baseline level). Note: Except for subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 hair loss, if the subject has undergone major surgery, the toxic reaction and/or complications caused by the surgical intervention must be fully recovered before starting treatment;
* Patients with multiple factors that affect oral medications (eg, inability to swallow, chronic diarrhea, and intestinal obstruction).
* Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage.
* Suffer from acute or chronic infectious diseases, such as hepatitis B, hepatitis C, tuberculosis, and HIV;
* Suffer from uncontrolled clinical symptoms or diseases of the heart, such as:(1) Heart failure above NYHA II; (2) Unstable angina pectoris; (3) Myocardial infarction occurred within 1 year; (4) Patients with clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention;
* Suffer from high blood pressure and cannot be well controlled by antihypertensive medication (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg);
* Live vaccines have been vaccinated within 4 weeks before the first use of the study drug.
* Active or previously documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea).
* Diagnosed as immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose >10mg/day prednisone or other equivalent therapeutic hormones), and still within 2 weeks before the first dose continue to use.
* Have a history of active pulmonary tuberculosis. In patients suspected of having active TB, examination of chest X-ray, sputum, and exclusion by clinical symptoms and signs are required.
* Has an active infection requiring systemic treatment.
* Previous history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis requiring hormone therapy, or any active interstitial lung disease with clinical evidence.
* Past history of clear neurological or psychiatric disorders.
* The investigator judged other situations not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-09-12 (Estimated); Primary Completion 2023-09-21 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | Time Frame: up to approximately 2 year
  Time from enrollment to first observation of progression (RECIST1.1) or date of death (from any cause)

SECONDARY OUTCOMES:
Objective response rate | Time Frame: up to approximately 1 year
  Proportion of patients with a complete or partial response as measured using RECIST 1.1 criteria
Overall Survival | Time Frame: up to approximately 2 year
  Time from enrollment until death due to any cause
incidence, type and severity of adverse events | Time Frame: up to approximately 2 year
  Descriptive statistics of safety will be presented using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0

IPD SHARING:
Plan to Share IPD: No